CLINICAL TRIAL: NCT00978341
Title: A Methodology Study to Assess the Ability of a Randomised, Double Blind, Placebo Controlled, Crossover Trial Design in Spinal Cord Injury Patients With Pain of Neuropathic Origin to Detect Improvement in Pain Endpoints Using Pregabalin as a Benchmark Compound
Brief Title: Study to Determine if a Reduction in Pain Can be Measured in Spinal Cord Injured Patients Using a New Study Design
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A0081141
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2009-11-09 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2010-01

CONDITIONS: Spinal Cord Injuries
Keywords: Clinical Trial Methodology study Neuropathic pain in Spinal cord injury patients Pain endpoints Crossover design
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin
- Placebo (Other)
  Interventions: Drug: Placebo for pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 150mg capsules BID for 7.5 days
  Arms: Pregabalin
Drug: Placebo for pregabalin — Placebo capsules BID for 7.5 days
  Arms: Placebo

SUMMARY:
The study is designed to assess if spinal cord injury patients have reduced pain after taking either pregabalin or placebo in a cross over design. Patients had either pain at the level of their injury or below the level of their injury.

DETAILED DESCRIPTION:
This methodology study was terminated on October 13, 2008 based on interim results for an exploratory, novel endpoint. The results of the primary analysis at the interim for N=12 patients showed results that generally favored pregabalin but were not statistically significant compared to placebo. Based on the estimated conditional power, this result is unlikely to change with full recruitment of N=24 patients and therefore the data monitoring committee recommended termination of the trial. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* subjects who are outpatients or inpatients
* written informed consent obtained (signed by the subject or the subject's legally acceptable representative)
* traumatic spinal cord injury of at least 1 year duration with a nonprogressive, i.e., chronic, stage of at least 6 months duration
* At-level neuropathic pain: spontaneous or evoked pain with neuropathic features (sharp, shooting, electric or burning pain sensation) in the region of sensory disturbance in a segmental pattern and located within two dermatomes above or below the level of spinal cord injury
* Below-level neuropathic pain: spontaneous or evoked pain with neuropathic features (sharp, shooting, electric or burning pain sensation) in the region of sensory disturbance located at least three dermatomes below the level of spinal cord injury

Exclusion Criteria:

* spinal cord injury (subjects with central pain and musculoskeletal pain must be able to make a distinction between the two)
* subjects who have previously not responded to 300 mg/day pregabalin: a non-responder is defined as a subject who has a reduction in pain score of less than 30% from baseline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Australia (4):
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Warrawong, New South Wales
  - Pfizer Investigational Site, Heidelberg, Victoria

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081141&StudyName=Study%20to%20determine%20if%20a%20reduction%20in%20pain%20can%20be%20measured%20in%20spinal%20cord%20injured%20patients%20using%20a%20new%20study%20design

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 4 study centers and participated in the study between 13 February 2007 and 01 October 2008.
Pre-assignment Details: Subjects completed a 1-2 week screening period to determine eligibility criteria prior to enrollment. Of 24 subjects screened, 15 subjects were enrolled into the study and randomized.
Groups:
- Pregabalin First Then Placebo: First Intervention Pregabalin Days 1-7: 150 mg twice a day (BID); Day 8: 150 mg in the morning. Second Intervention Placebo Days 1-7: twice a day (BID); Day 8: 1 dose in the morning.
- Placebo First Then Pregabalin: First Intervention Placebo Days 1-7: twice a day (BID); Day 8: 1 dose in the morning. Second Intervention Pregabalin: Days 1-7: 150 mg twice a day (BID); Day 8: 150 mg in the morning.
Period: First Intervention
Arm/Group | Pregabalin First Then Placebo | Placebo First Then Pregabalin
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | Pregabalin First Then Placebo | Placebo First Then Pregabalin
Started | 8 | 7
Completed | 7 | 7
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Second Intervention
Arm/Group | Pregabalin First Then Placebo | Placebo First Then Pregabalin
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Pregabalin: Days 1-7: 150 mg twice a day (BID); Day 8: 150 mg in the morning; and Placebo: Days 1-7: twice a day (BID); Day 8: 1 dose in the morning.
Arm/Group | All Subjects
Number analyzed (Participants) | 15
Age, Customized [Number; unit: participants]
  18-44 years | 5
  45-64 years | 7
  >= 65 years | 3
Sex/Gender, Customized [Number; unit: gender]
  Female | 2
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Present Pain Intensity Score
Description: Present pain intensity score: 0-10 numeric rating scale (NRS), 0 (no pain) to 10 (worst possible pain).
Time Frame: Day 1: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours (post-dose); Day 8: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours (post-dose)
Population: Full analysis set (FAS): those subjects who completed both periods of the study. Combined results for At-level and Below-level neuropathic pain; At-level: located within 2 dermatomes above or below the level of spinal cord injury; Below-level: located at least 3 dermatomes below the level of spinal cord injury.
Measure: Mean (Standard Deviation); unit: scores on scale
Groups:
- Pregabalin: Days 1-7: 150 mg twice a day (BID); Day 8: 150 mg in the morning.
- Placebo: Days 1-7: twice a day (BID); Day 8: 1 dose in the morning
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 15 | 14
scores on scale
  Day 1: pre-dose (n=15, 14) | 5.3 (2.76) | 4.9 (2.91)
  Day 1: 0.5 hours post-dose (n=15, 14) | 5.1 (2.46) | 4.6 (3.03)
  Day 1: 1 hours post-dose (n=15, 14) | 4.6 (2.82) | 4.7 (2.55)
  Day 1: 2 hours post-dose (n=15, 14) | 4.3 (2.64) | 4.7 (2.64)
  Day 1: 3 hours post-dose (n=15, 14) | 4.3 (2.82) | 4.7 (2.73)
  Day 1: 4 hours post-dose (n=15, 14) | 4.1 (2.79) | 4.6 (2.98)
  Day 1: 5 hours post-dose (n=15, 14) | 3.9 (3.01) | 4.9 (3.02)
  Day 1: 6 hours post-dose (n=15, 14) | 3.9 (2.89) | 5.1 (2.91)
  Day 1: 8 hours post-dose (n=15, 14) | 4.3 (2.91) | 5.1 (2.57)
  Day 1: 10 hours post-dose (n=14, 14) | 4.1 (3.03) | 5.3 (2.81)
  Day 1: 12 hours post-dose (n=14, 14) | 4.1 (3.17) | 5.4 (2.68)
  Day 8: pre-dose (n=13, 14) | 4.7 (2.53) | 5.4 (2.62)
  Day 8: 0.5 hours post-dose (n=13, 14) | 4.5 (2.33) | 5.0 (2.57)
  Day 8: 1 hour post-dose (n=13, 14) | 4.0 (2.71) | 4.9 (2.60)
  Day 8: 2 hours post-dose (n=13, 14) | 4.6 (2.50) | 4.6 (2.38)
  Day 8: 3 hours post-dose (n=15, 14) | 4.9 (2.22) | 4.7 (2.52)
  Day 8: 4 hours post-dose (n=15, 14) | 4.9 (2.28) | 4.9 (2.53)
  Day 8: 5 hours post-dose (n=15, 14) | 4.8 (2.40) | 4.9 (2.63)
  Day 8: 6 hours post-dose (n=15, 14) | 4.4 (2.38) | 5.2 (2.72)
  Day 8: 8 hours post-dose (n=15, 13) | 4.7 (2.63) | 5.3 (2.90)
  Day 8: 10 hours post-dose (n=15, 13) | 4.9 (2.37) | 5.2 (2.85)
  Day 8: 12 hours post-dose (n=15, 13) | 4.7 (2.16) | 5.2 (2.65)
  Day 8: 24 hours post-dose (n=15, 14) | 5.0 (2.36) | 5.4 (2.71)
  Day 8: 36 hours post-dose (n=15, 13) | 6.1 (2.74) | 5.7 (2.56)
  Day 8: 48 hours post-dose (n=15, 14) | 6.1 (2.31) | 5.8 (2.81)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 1: 0.5 hours post-dose; Test type: Superiority or Other; p = 0.6797, ANOVA; Mean Difference (Final Values) = 0.20, 95% CI [-0.83 to 1.22], Standard Error of Mean 0.462
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 1: 1 hour post-dose; Test type: Superiority or Other; p = 0.4811, ANOVA; Mean Difference (Final Values) = -0.38, 95% CI [-1.54 to 0.77], Standard Error of Mean 0.528
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 1: 2 hours post-dose; Test type: Superiority or Other; p = 0.1693, ANOVA; Mean Difference (Final Values) = -0.67, 95% CI [-1.67 to 0.33], Standard Error of Mean 0.454
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline) , Day 1: 3 hours post-dose; Test type: Superiority or Other; p = 0.4034, ANOVA; Mean Difference (Final Values) = -0.45, 95% CI [-1.78 to 0.87], Standard Error of Mean 0.487
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 1: 4 hours post-dose; Test type: Superiority or Other; p = 0.1935, ANOVA; Mean Difference (Final Values) = -0.93, 95% CI [-2.36 to 0.50], Standard Error of Mean 0.694
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 1: 5 hours post-dose; Test type: Superiority or Other; p = 0.0694, ANOVA; Mean Difference (Final Values) = -1.36, 95% CI [-2.83 to 0.12], Standard Error of Mean 0.715
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 1: 6 hours post-dose; Test type: Superiority or Other; p = 0.0396, ANOVA; Mean Difference (Final Values) = -1.55, 95% CI [-3.02 to -0.08], Standard Error of Mean 0.713
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 1: 8 hours post-dose; Test type: Superiority or Other; p = 0.1531, ANOVA; Mean Difference (Final Values) = -0.51, 95% CI [-1.25 to 0.24], Standard Error of Mean 0.319
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 1: 10 hours post-dose; Test type: Superiority or Other; p = 0.0951, ANOVA; Mean Difference (Final Values) = -1.25, 95% CI [-2.79 to 0.29], Standard Error of Mean 0.637
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 1: 12 hours post-dose; Test type: Superiority or Other; p = 0.0614, ANOVA; Mean Difference (Final Values) = -1.38, 95% CI [-2.84 to 0.09], Standard Error of Mean 0.615
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: pre-dose; Test type: Superiority or Other; p = 0.1946, ANOVA; Mean Difference (Final Values) = -0.87, 95% CI [-2.29 to 0.54], Standard Error of Mean 0.619
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 0.5 hours post-dose; Test type: Superiority or Other; p = 0.2843, ANOVA; Mean Difference (Final Values) = -0.68, 95% CI [-2.20 to 0.84], Standard Error of Mean 0.553
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 1 hour post-dose; Test type: Superiority or Other; p = 0.2150, ANOVA; Mean Difference (Final Values) = -1.05, 95% CI [-2.75 to 0.65], Standard Error of Mean 0.820
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 2 hours post-dose; Test type: Superiority or Other; p = 0.9601, ANOVA; Mean Difference (Final Values) = -0.01, 95% CI [-0.44 to 0.42], Standard Error of Mean 0.189
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Difference from placebo (including baseline), Day 8: 3 hours post-dose; Test type: Superiority or Other; p = 0.8670, ANOVA; Mean Difference (Final Values) = 0.05, 95% CI [-0.64 to 0.74], Standard Error of Mean 0.311
Statistical Analysis 16: Comparison: Pregabalin vs Placebo; Difference from placebo (including baseline), Day 8: 4 hours post-dose; Test type: Superiority or Other; p = 0.9024, ANOVA; Mean Difference (Final Values) = -0.05, 95% CI [-0.94 to 0.84], Standard Error of Mean 0.393
Statistical Analysis 17: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 5 hours post-dose; Test type: Superiority or Other; p = 0.9708, ANOVA; Mean Difference (Final Values) = -0.01, 95% CI [-0.67 to 0.65], Standard Error of Mean 0.293
Statistical Analysis 18: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 6 hours post-dose; Test type: Superiority or Other; p = 0.1078, ANOVA; Mean Difference (Final Values) = -0.71, 95% CI [-1.62 to 0.19], Standard Error of Mean 0.395
Statistical Analysis 19: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 8 hours post-dose; Test type: Superiority or Other; p = 0.4460, ANOVA; Mean Difference (Final Values) = -0.33, 95% CI [-1.28 to 0.61], Standard Error of Mean 0.419
Statistical Analysis 20: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 10 hours post-dose; Test type: Superiority or Other; p = 0.5266, ANOVA; Mean Difference (Final Values) = -0.26, 95% CI [-1.13 to 0.62], Standard Error of Mean 0.394
Statistical Analysis 21: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 12 hours post-dose; Test type: Superiority or Other; p = 0.0290, ANOVA; Mean Difference (Final Values) = -0.69, 95% CI [-1.29 to -0.08], Standard Error of Mean 0.273
Statistical Analysis 22: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 24 hours post-dose; Test type: Superiority or Other; p = 0.1830, ANOVA; Mean Difference (Final Values) = -0.78, 95% CI [-2.01 to 0.45], Standard Error of Mean 0.531
Statistical Analysis 23: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 36 hours post-dose; Test type: Superiority or Other; p = 0.9884, ANOVA; Mean Difference (Final Values) = 0.01, 95% CI [-0.90 to 0.91], Standard Error of Mean 0.406
Statistical Analysis 24: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline), Day 8: 48 hours post-dose; Test type: Superiority or Other; p = 0.8082, ANOVA; Mean Difference (Final Values) = -0.09, 95% CI [-0.87 to 0.69], Standard Error of Mean 0.354

2. Secondary Outcome: Daily Pain Score
Description: Daily Pain Score: Day 1 pain intensity over past 24 hours recorded on waking every morning. 0-10 numeric rating scale (NRS): 0 (no pain) to 10 (worst possible pain).
Time Frame: Predose: Daily from 7 days before Visit 2 (start of Intervention 1) until the morning of Visit 5 (end of Intervention 2)
Population: FAS; Combined results for At-level and Below-level of spinal cord injury.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 15 | 14
scores on scale
  Day 1 (n=15, 13) | 6.2 (1.78) | 6.3 (2.06)
  Day 2 (n=15, 14) | 4.4 (2.67) | 5.4 (2.47)
  Day 3 (n=15, 14) | 4.1 (2.49) | 5.1 (2.35)
  Day 4 (n=15, 14) | 4.2 (2.51) | 5.0 (2.35)
  Day 5 (n= 15, 14) | 4.5 (2.67) | 5.1 (2.37)
  Day 6 (n=15, 14) | 3.7 (2.60) | 4.9 (2.30)
  Day 7 (n=15, 14) | 4.0 (2.70) | 4.9 (2.54)
  Day 8 (n=14, 14) | 4.0 (2.35) | 5.6 (2.47)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Difference from placebo (including baseline); Day 2. Combined analysis: values for the two patient groups were analyzed together using ANOVA and/or mixed models; Test type: Superiority or Other; p = 0.2101, ANOVA; Mean Difference (Final Values) = -0.92, 95% CI [-2.39 to 0.55], Standard Error of Mean 0.714
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Difference from placebo (including baseline); Day 3; Test type: Superiority or Other; p = 0.1065, ANOVA; Mean Difference (Final Values) = -1.04, 95% CI [-2.33 to 0.24], Standard Error of Mean 0.623
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Difference from placebo (including baseline); Day 4; Test type: Superiority or Other; p = 0.0697, ANOVA; Mean Difference (Final Values) = -0.53, 95% CI [-1.11 to 0.05], Standard Error of Mean 0.254
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Difference from placebo; Day 5; Test type: Superiority or Other; p = 0.4589, ANOVA; Mean Difference (Final Values) = -0.49, 95% CI [-1.83 to 0.85], Standard Error of Mean 0.650
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Difference from placebo; Day 6; Test type: Superiority or Other; p = 0.1326, ANOVA; Mean Difference (Final Values) = -1.16, 95% CI [-2.69 to 0.38], Standard Error of Mean 0.742
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Difference from placebo (including baseline); Day 7; Test type: Superiority or Other; p = 0.2820, ANOVA; Mean Difference (Final Values) = -0.78, 95% CI [-2.45 to 0.90], Standard Error of Mean 0.638
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Difference from placebo (including baseline); Day 8; Test type: Superiority or Other; p = 0.0108, ANOVA; Mean Difference (Final Values) = -1.33, 95% CI [-2.21 to -0.44], Standard Error of Mean 0.356

3. Secondary Outcome: Dynamic Allodynia Area
Description: Area of dynamic allodynia was assessed using a brush (SENSElab Brush 05; velocity approximately 20 millimeters per second [mm/s]) by stimulating along a pattern of 8 radial spokes. Stimulation was started from the non-painful perimetry. Subjects were asked to report change in sensation from non-painful to painful and the spot was marked onto the skin. The area of dynamic allodynia was determined from these 8 distances by calculating the area of an octagon (in centimeter squared [cm2]).
Time Frame: Screening, Days 1 & 8: 0 (pre-dose) & 4 hours post-dose,
Population: FAS; Combined results for At-level and Below-level of spinal cord injury.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 15 | 14
cm2
  Day 1: pre-dose (n=14, 14) | 95.8 (108.1) | 81.6 (111.2)
  Day 1: 4 hours post-dose (n=15, 13) | 63.0 (78.54) | 50.9 (78.64)
  Day 8: pre-dose (n=12, 14) | 48.4 (92.07) | 68.4 (83.53)
  Day 8: 4 hours post-dose (n=15, 13) | 50.5 (83.72) | 68.0 (91.41)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Difference from placebo; Day 1: 4 hours post-dose (including Baseline); Test type: Superiority or Other; p = 0.9068, ANOVA; Mean Difference (Final Values) = -2.26, 95% CI [-41.78 to 37.27], Standard Error of Mean 19.060
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Difference from placebo; Day 8: pre-dose (including Baseline); Test type: Superiority or Other; p = 0.7807, ANOVA; Mean Difference (Final Values) = 4.52, 95% CI [-30.53 to 39.57], Standard Error of Mean 15.813
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Difference from placebo; Day 8: 4 hours post-dose (including Baseline); Test type: Superiority or Other; p = 0.2293, ANOVA; Mean Difference (Final Values) = -22.51, 95% CI [-61.79 to 16.78], Standard Error of Mean 17.526

4. Secondary Outcome: Dynamic Allodynia Pain Score
Description: Five strokes (each approx. 6 centimeters [cm] long) were applied with a standardized brush (SENSELab Brush 05) across the painful site (and a control site) at a constant velocity (20 millimeters per second [mm/sec]). Pain in response to brush stimulation of the allodynic area was recorded using an 11-point numeric rating scale from 0 (no pain) to 10 (worst possible pain). Patients were asked to give a pain rating after each brush stroke. A painful sensation was considered as representing brush allodynia.
Time Frame: Screening, Days 1 & 8: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, and 6 hours post-dose
Population: FAS; Combined results for At-level and Below-level of spinal cord injury.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 15 | 14
scores on scale
  Day 1: pre-dose (n=14, 13) | 2.2 (2.99) | 2.1 (3.33)
  Day 1: 0.5 hours post-dose (n=10, 8) | 2.8 (3.14) | 1.9 (3.35)
  Day 1: 1 hour post-dose (n=10, 8) | 2.3 (2.83) | 1.8 (3.15)
  Day 1: 2 hours post-dose (n=10, 8) | 2.5 (3.09) | 1.7 (2.67)
  Day 1: 3 hours post-dose (n=10, 8) | 2.3 (2.94) | 2.3 (2.98)
  Day 1: 4 hours post-dose (n=15, 13) | 1.5 (2.63) | 1.2 (2.28)
  Day 1: 5 hours post-dose (n=10, 8) | 2.2 (2.95) | 1.9 (2.70)
  Day 1: 6 hours post-dose (n=10, 8) | 2.1 (2.80) | 1.9 (2.75)
  Day 8: pre-dose (n=11, 12) | 1.9 (2.93) | 2.0 (2.97)
  Day 8: 0.5 hours post-dose (n=7, 8) | 1.7 (2.74) | 1.7 (2.66)
  Day 8: 1 hour post-dose (n=7, 8) | 1.6 (2.66) | 1.4 (2.58)
  Day 8: 2 hours post-dose (n=7, 8) | 1.9 (2.93) | 1.5 (2.43)
  Day 8: 3 hours post-dose (n=9, 8) | 1.7 (2.45) | 1.6 (2.51)
  Day 8: 4 hours post-dose (n=14, 13) | 1.0 (1.99) | 0.9 (1.99)
  Day 8: 5 hours post-dose (n=9, 8) | 1.9 (2.83) | 1.5 (2.40)
  Day 8: 6 hours post-dose (n=9, 8) | 1.9 (3.05) | 1.5 (2.57)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 0.5 hours post-dose; Test type: Superiority or Other; p = 0.3774, ANOVA; Mean Difference (Final Values) = 0.36, 95% CI [-0.54 to 1.27], Standard Error of Mean 0.386
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 1 hour post-dose; Test type: Superiority or Other; p = 0.4153, ANOVA; Mean Difference (Final Values) = 0.19, 95% CI [-0.33 to 0.70], Standard Error of Mean 0.215
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 2 hours post-dose; Test type: Superiority or Other; p = 0.1470, ANOVA; Mean Difference (Final Values) = 0.48, 95% CI [-0.23 to 1.20]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 3 hours post-dose; Test type: Superiority or Other; p = 0.1862, ANOVA; Mean Difference (Final Values) = -0.45, 95% CI [-1.18 to 0.29], Standard Error of Mean 0.300
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 4 hours post-dose; Test type: Superiority or Other; p = 0.8321, ANOVA; Mean Difference (Final Values) = 0.05, 95% CI [-0.45 to 0.55], Standard Error of Mean 0.220
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 5 hours post-dose; Test type: Superiority or Other; p = 0.4251, ANOVA; Mean Difference (Final Values) = 0.23, 95% CI [-0.42 to 0.88], Standard Error of Mean 0.269
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 6 hours post-dose; Test type: Superiority or Other; p = 0.6394, ANOVA; Mean Difference (Final Values) = 0.13, 95% CI [-0.53 to 0.80], Standard Error of Mean 0.269
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: pre-dose; Test type: Superiority or Other; p = 0.9964, ANOVA; Mean Difference (Final Values) = 0.00, 95% CI [-0.68 to 0.68], Standard Error of Mean 0.302
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 0.5 hours post-dose; Test type: Superiority or Other; p = 0.3638, ANOVA; Mean Difference (Final Values) = 0.32, 95% CI [-0.47 to 1.11], Standard Error of Mean 0.324
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 1 hour post-dose; Test type: Superiority or Other; p = 0.1202, ANOVA; Mean Difference (Final Values) = 0.42, 95% CI [-0.15 to 0.99], Standard Error of Mean 0.223
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 2 hours post-dose; Test type: Superiority or Other; p = 0.1204, ANOVA; Mean Difference (Final Values) = 0.60, 95% CI [-0.19 to 1.39], Standard Error of Mean 0.355
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 3 hours post-dose; Test type: Superiority or Other; p = 0.4213, ANOVA; Mean Difference (Final Values) = 0.25, 95% CI [-0.44 to 0.93], Standard Error of Mean 0.289
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 4 hours post-dose; Test type: Superiority or Other; p = 0.6028, ANOVA; Mean Difference (Final Values) = 0.11, 95% CI [-0.34 to 0.56], Standard Error of Mean 0.205
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 5 hours post-dose; Test type: Superiority or Other; p = 0.3624, ANOVA; Mean Difference (Final Values) = 0.48, 95% CI [-0.68 to 1.64], Standard Error of Mean 0.491
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 6 hours post-dose; Test type: Superiority or Other; p = 0.3163, ANOVA; Mean Difference (Final Values) = 0.48, 95% CI [-0.52 to 1.49], Standard Error of Mean 0.461

5. Secondary Outcome: Punctate Allodynia Area
Description: Area of punctate allodynia was determined using a von Frey filament (OptiHair2). Stimulation was started from the non-painful perimetry and repeated along a pattern of 8 radial spokes. With a movement along each spoke at steps of 5 millimeters (mm), the subjects reported sensation changes from non-painful to painful and the spot was marked on the skin. The area of punctate allodynia was determined from these 8 distances by calculating the area of an octagon (in square centimeter(s)[cm2]).
Time Frame: Screening, Days 1 & 8: 0 (pre-dose) and 4 hours post-dose
Population: FAS; combined results for At-level and Below-level spinal cord injury.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 15 | 14
cm2
  Day 1: pre-dose (n=15, 14) | 75.6 (113.3) | 65.1 (104.8)
  Day 1: 4 hours post-dose (n=15, 13) | 68.7 (112.6) | 54.1 (91.21)
  Day 8: pre-dose (n=13, 14) | 53.1 (102.2) | 45.9 (74.32)
  Day 8: 4 hours post-dose (n=15, 13) | 70.8 (106.3) | 46.7 (80.73)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1; Test type: Superiority or Other; p = 0.5919, ANOVA; Mean Difference (Final Values) = 5.39, 95% CI [-16.26 to 27.04], Standard Error of Mean 9.738
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: pre-dose; Test type: Superiority or Other; p = 0.3981, ANOVA; Mean Difference (Final Values) = 12.58, 95% CI [-17.70 to 42.87], Standard Error of Mean 14.603
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 4 hours post-dose; Test type: Superiority or Other; p = 0.8314, ANOVA; Mean Difference (Final Values) = 2.64, 95% CI [-24.00 to 29.28], Standard Error of Mean 12.123

6. Secondary Outcome: Mechanical Pain Sensitivity Stimulus-Response Function
Description: Mechanical pain sensitivity stimulus response function was assessed at the control and painful sites using calibrated von Frey monofilaments and the SENSElab brush. Seven different von Frey monofilaments (8 -512 milliNewtons [mN], force increases by a factor of two from filament to filament) and the brush were applied in a predetermined pseudo-random order. Pain rating for each stimulus: 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Screening, Days 1 & 8: 0 (pre-dose), & 2, 4, and 6 hours post-dose
Population: FAS; combined results for At-level and Below-level of spinal cord injury.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 14 | 14
scores on scale
  Day 1: pre-dose (n=14, 14) | 0.8 (0.78) | 0.9 (0.73)
  Day 1: 2 hours post-dose (n=14, 14) | 0.7 (0.58) | 0.8 (0.65)
  Day 1: 4 hours post-dose (n=14, 14) | 0.7 (0.64) | 0.8 (0.65)
  Day 1: 6 hours post-dose (n=14, 14) | 0.8 (0.61) | 0.9 (0.68)
  Day 8: pre-dose (n=13, 14) | 0.7 (0.61) | 0.8 (0.64)
  Day 8: 2 hours post-dose (=13, 14) | 0.7 (0.50) | 0.8 (0.66)
  Day 8: 4 hours post-dose (n=15, 13) | 0.7 (0.65) | 0.7 (0.62)
  Day 8: 6 hours post-dose (n=15, 13) | 0.8 (0.67) | 0.7 (0.59)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 2 hours post-dose; Test type: Superiority or Other; p = 0.7569, ANOVA; Mean Difference (Final Values) = -0.02, 95% CI [-0.14 to 0.10], Standard Error of Mean 0.054
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 4 hours post-dose; Test type: Superiority or Other; p = 0.4814, ANOVA; Mean Difference (Final Values) = -0.07, 95% CI [-0.26 to 0.13], Standard Error of Mean 0.090
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 1: 6 hours post-dose; Test type: Superiority or Other; p = 0.6222, ANOVA; Mean Difference (Final Values) = -0.07, 95% CI [-0.37 to 0.23], Standard Error of Mean 0.143
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: pre-dose; Test type: Superiority or Other; p = 0.3035, ANOVA; Mean Difference (Final Values) = -0.12, 95% CI [-0.35 to 0.12], Standard Error of Mean 0.113
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 2 hours post-dose; Test type: Superiority or Other; p = 0.1881, ANOVA; Mean Difference (Final Values) = -0.17, 95% CI [-0.42 to 0.09], Standard Error of Mean 0.122
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 4 hours post-dose; Test type: Superiority or Other; p = 0.3159, ANOVA; Mean Difference (Final Values) = 0.08, 95% CI [-0.09 to 0.24], Standard Error of Mean 0.072
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Difference from placebo (including Baseline); Day 8: 6 hours post-dose; Test type: Superiority or Other; p = 0.8203, ANOVA; Mean Difference (Final Values) = 0.02, 95% CI [-0.22 to 0.27], Standard Error of Mean 0.103

7. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI)
Description: NPSI: subject rated questionnaire to evaluate 5 dimensions of neuropathic pain (dimensions: burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia). Includes 10 descriptors ranging from 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. Questionnaire generates a score in each relevant dimension. Total score is calculated as the sum of scores of the 10 descriptors, range: 0-100. Higher score indicates greater intensity of pain.
Time Frame: Prior to morning dosing on Day 1 and prior to discharge on Day 8 for each period.
Population: FAS; Combined results for At-level and Below-level of spinal cord injury.
Measure: Median (Inter-Quartile Range); unit: scores on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 15 | 14
scores on scale
  Category 1 Day 1 (n=15, 14) | 6.0 [3.0 to 7.0] | 6.0 [0.0 to 7.0]
  Category 1: Day 8 (n=12, 11) | 5.5 [1.5 to 7.0] | 6.0 [0.0 to 7.0]
  Category 2: Day 1 (n=15, 14) | 3.0 [1.0 to 5.0] | 2.5 [1.0 to 4.0]
  Category 2: Day 8 (n=12, 11) | 2.5 [1.5 to 3.3] | 3.0 [2.0 to 4.5]
  Category 3: Day 1 (n=15, 14) | 1.5 [0.0 to 5.0] | 3.3 [1.0 to 5.0]
  Category 3: Day 8 (n=12, 11) | 1.8 [0.0 to 3.5] | 2.0 [0.0 to 5.0]
  Category 4: Day 1 (n=15, 14) | 1.7 [0.0 to 6.0] | 0.3 [0.0 to 3.3]
  Category 4: Day 8 (n=12, 11) | 2.7 [0.8 to 4.7] | 0.0 [0.0 to 4.0]
  Category 5: Day 1 (n=15, 14) | 5.0 [0.0 to 7.0] | 5.0 [1.5 to 7.0]
  Category 5: Day 8 (n=12, 11) | 3.5 [1.5 to 5.5] | 5.0 [2.0 to 6.0]
  Total: Day 1 (n=15, 14) | 32 [14.0 to 48.0] | 27 [21.0 to 42.0]
  Total: Day 8 (n=12, 11) | 22 [18.5 to 51.5] | 24 [20.0 to 46.0]

8. Secondary Outcome: Pharmacokinetic Evaluations of Pregabalin
Description: Pharmacokinetic (PK) results are not presented in this report due to early termination of the trial. Pregabalin PK was not measured as there was incomplete data to conduct pharmacokinetic/pharmacodynamic analyses.
Time Frame: Day 1: 0 (pre-dose), 0.5, 1, 2, and 6 hours post-dose; Day 8: 0 (pre-dose), 1, 4, & 6 hours post-dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/14
Other Adverse Events (participants affected / at risk) | 12/15 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=15) | Placebo (N=14)
Urinary tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=15) | Placebo (N=14)
Palpitations (Cardiac disorders) | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 1
Eye pain (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Catheter related complication (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Feeling drunk (General disorders) | 2 | 0
Feeling hot (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 1
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1
Muscle spasticity (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 5 | 2
Tension headache (Nervous system disorders) | 1 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other